CLINICAL TRIAL: NCT06073587
Title: CARDIO-TTRansform ION-682884-CS2-Scintigraphy Sub-study
Brief Title: The CARDIO-TTRansform Scintigraphy Sub-study
Status: Active, not recruiting | Type: Observational
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: ION-682884-CS2-Scintigraphy; 2019-002835-27 (EudraCT Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Transthyretin-Mediated Amyloid Cardiomyopathy (ATTR-CM)
Keywords: TTR; Amyloidosis; Cardiomyopathy
MeSH Terms: conditions — Amyloidosis; Cardiomyopathies | interventions — Ventilation-Perfusion Scan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ION-682884-CS2 Scintigraphy Subset: Participants randomized in ION-682884-CS2 (NCT04136171) study to receive either eplontersen or placebo with baseline scintigraphy scan with planar and single-photon emission computerized tomography (SPECT) or SPECT with computed tomography (SPECT/CT) images will undergo an optional scintigraphy scan at Weeks 25 or 37, Week 97, and an additional scan at Week 140.
  Interventions: Diagnostic Test: Scintigraphy scan

INTERVENTIONS:
Diagnostic Test: Scintigraphy scan — Scans will be performed as specified in the arm description.

SUMMARY:
The purpose of this study is to examine the changes in amyloid myocardial burden in a subset of the population participating in the ION682884-CS2 (NCT04136171) study, up to 150 participants, after treatment with eplontersen or placebo based on scintigraphy scans performed at Week 140 using the Perugini grade score method.

DETAILED DESCRIPTION:
Participants who were randomized in Study ION-682884-CS2 (NCT04136171) and have had a baseline scintigraphy scan will be offered the opportunity to participate in this sub-study which involves optional scintigraphy scans.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been properly randomized into the ION-682884-CS2 study (NCT04136171) and should have had a baseline scintigraphy scan (99mTc-DPD, 99mTc- PYP, and 99mTc-HMDP) within 12 months prior to screening for ION-682884-CS2 with planar and SPECT or SPECT/CT images that can be read by the central reader.

Exclusion criteria:

* Must not meet any of the exclusion criteria of the study protocol ION-682884-CS2 (NCT04136171).
* Must not have weight or body girth that exceeds the limits of the equipment specifications.
* Should not have any previously reported hypersensitivity reaction to Technetium-99m.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were randomized in Study ION-682884-CS2 (NCT04136171) and who signed informed consent for the Scintigraphy sub-study will participate in this sub-study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes From Baseline in Perugini Grading Score From Scintigraphy Scan Images at Week 140 | Baseline up to Week 140
  The Perugini grading scale visually compares tracer uptake in the myocardium and ribs following injection of the bone tracers (99mTc-DPD, 99mTc-Pyrophosphate [PYP], or 99mTc-HMDP). The scale includes 4 grade classifications: Grade 0- no cardiac uptake and normal rib uptake, Grade 1- cardiac uptake which is less than rib uptake, Grade 2- cardiac uptake with intensity similar rib uptake, and Grade 3- cardiac uptake greater than rib uptake with mild or absent rib uptake. Visual scores of 2 or greater are classified as ATTR-positive and less than 2 are interpreted as ATTR-negative.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Columbia University Irving Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
- Hospital Universitario Puerta de Hierro, Majadahonda, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: CARDIO-TTRansform Website — https://www.cardio-ttransform.com/